CLINICAL TRIAL: NCT06882837
Title: Body Weight Awareness and SUpport for Mums During Pregnancy (BUMP2.0): a Feasibility Study
Brief Title: BUMP2.0 Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, DrMoschoMichalopoulou, Post-doctoral Researcher - Behavioural Scientist, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R95714/RE001
Record Dates: First submitted 2025-02-17; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Weight Gain During Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BUMP app (Experimental)
  Interventions: Behavioral: BUMP app
- Usual care (No Intervention): No intervention

INTERVENTIONS:
Behavioral: BUMP app — Participants in the experimental group will have access to the BUMP app, which aims to support them to control the amount and rate of weight gain during pregnancy, from baseline (early or mid-pregnancy) until they give birth. The app will prompt participants to regularly self-monitor their weight gain during pregnancy, and will provide access to a weight gain chart for tracking. Participants will receive feedback notifications about their weight gain trajectory, and will have access to information and tips on weight management during pregnancy.
  Arms: BUMP app

SUMMARY:
Most women in the UK gain more weight than recommended during pregnancy, which puts them and their babies at risk of medical complications. Studies which have interviewed women during pregnancy have shown that they recognise that controlling their weight is important, but this is rarely discussed with their clinical team. Some women reported they expected to be weighed during pregnancy, and that regular weighing should be part of routine antenatal care, but it is not. Trials which have trained midwives to regularly weigh women or to ask women to regularly weigh themselves, have not shown beneficial effects on gestational weight gain. However, these trials were either small, or reported low protocol adherence, or did not offer adequate feedback and advice in response to weight gain. A few programmes to manage weight during pregnancy have been effective, but were costly and burdensome for women. Regular self-weighing has been shown to be an effective strategy for weight control outside of pregnancy, and if it can be enacted in pregnancy and help manage weight gain, it could improve health outcomes for women and their babies.

The investigators have developed a mobile app to support women to weigh themselves regularly during pregnancy and track their weight gain, to provide feedback on whether weight gain is within, higher, or lower than recommended ranges, and to signpost to resources on weight management during pregnancy. The trial aims to test if it is possible to motivate participants to regularly weigh themselves during pregnancy and how well they engage with the app from early or mid-pregnancy until delivery. The investigators will also examine whether the processes of the study run as planned, whether there is an indication of an impact of the programme on gestational weight gain compared to a control group, and will explore participants' experiences of using the app through optional qualitative interviews. If feasible, after completion of this study, the next step will be a bigger trial to investigate whether this app-based programme is effective in helping women manage their weight gain and improve health outcomes during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at <20 weeks' gestation
* 18 years of age or above
* Singleton pregnancy
* 18 years of age or above
* Able to access the internet with a smartphone and/or tablet
* Have access to weighing scales
* Able to communicate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants in the BUMP app group who log their weight on at least half of all weeks of their participation | From randomization which can happen any time between the start of pregnancy and 20 weeks of pregnancy, until the end of the study for each participant, which is the date on which a participant gives birth, usually at 40-42 weeks of pregnancy.
Percentage of participants in the BUMP app group who spontaneously log a weight measurement into the app at later stages of pregnancy | Late stages of pregnancy, defined as the time frame between 34 weeks of pregnancy and the date on which a participant gives birth usually at 40-42 weeks of pregnancy.
Overall retention rate at study follow-up | Late stages of pregnancy, defined as the time frame between 34 weeks of pregnancy and the date on which a participant gives birth usually at 40-42 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuffield Department of Primary Care Health Sciences, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided